CLINICAL TRIAL: NCT05679167
Title: Digital Training Interventions for Low Back Pain - RCT With Longitudinal Evaluation of Clinical Outcome Measures and MRI Examinations
Brief Title: Digital Training Interventions for Low Back Pain
Acronym: DigiLum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Ninni Sernert, Professor, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vastra Gotaland
Record Dates: First submitted 2022-11-10; First posted 2023-01-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
Keywords: MRI; Physiotherapy; Supervised digital training
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Three ongoing different treatments at the same time
Masking Description: Both patients and physiotherapists know what intervention group they were randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised digital training: core stability (Active Comparator): The patients will be identified at the primary health center and after fulfilling the inclusion criteria and all baseline examination are completed the patients will be randomized. In group 1 the patients will attend supervised digital training with focus on core stability
  Interventions: Behavioral: Supervised digital training with focus on aerobic exercise; Behavioral: Non-supervised daily physical activity
- Supervised digital training: aerobic exercise (Active Comparator): The patients will be identified at the primary health center and after fulfilling the inclusion criteria and all baseline examination are completed the patients will be randomized. In group 2 the patients will attend supervised digital training with focus on aerobic exercise
  Interventions: Behavioral: Supervised digital training with focus on core stability; Behavioral: Non-supervised daily physical activity
- Non-supervised daily physical activity (Active Comparator): The patients will be identified at the primary health center and after fulfilling the inclusion criteria and all baseline examination are completed the patients will be randomized. In group 3 will start a daily physical activity program, with regular support from a physiotherapist.
  Interventions: Behavioral: Supervised digital training with focus on core stability; Behavioral: Supervised digital training with focus on aerobic exercise

INTERVENTIONS:
Behavioral: Supervised digital training with focus on core stability — After randomization, Group 1 will be digitally supervised by experienced physiotherapist.
  Arms: Non-supervised daily physical activity; Supervised digital training: aerobic exercise
Behavioral: Supervised digital training with focus on aerobic exercise — After randomization Group 2 will be digitally supervised by experienced physiotherapist.
  Arms: Non-supervised daily physical activity; Supervised digital training: core stability
Behavioral: Non-supervised daily physical activity — After randomization Group 3 will receive training instruction regarding daily physical activity.
  Arms: Supervised digital training: aerobic exercise; Supervised digital training: core stability

SUMMARY:
The patients will be clinically examined, as well as evaluated with Patient Reported Outcome Measures (PROMs) and Magnet Resonance Imaging (MRI) at baseline and at follow-ups.

DETAILED DESCRIPTION:
The overall aim is to evaluate two different types of digital training interventions supervised by physiotherapists compared to daily physical activity in terms of clinical, imaging-based and patient-reported outcome in patients with low back pain. Furthermore, to evaluate whether new diagnostic MRI methods can identify longitudinal spine tissue changes and to analyse if there is an exercise-related difference.

Patients seeking primary health care for lower back pain will be randomized to three groups. The patients will be clinically examined, assessed with Magnet Resonance Imaging (MRI) and Patient Reported Outcome Measures (PROMs) will be evaluated at baseline and at follow-ups.

A detailed description of the study protocol, see attached document.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain> 3 months
* Age 18-50 years
* Access to computer/tablet/mobile phone

Exclusion Criteria:

* Inadequate Swedish as the language is an obstacle to be able to fully understand written and oral information regarding the project and to follow training instructions
* Other ongoing treatment/exercise for their low back pain
* Patients with radiating leg pain and neurological symptoms where herniated discs are suspected
* Previous back/neck surgery
* Pregnancy
* Diagnosed systematic diseases engaging the spine as rheumatoid arthritis, ankylosing spondylitis
* Factors that prevent an MRI examination, such as claustrophobia, metal implants, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-reported pain | 6 months compared to baseline
  Visual Analog Scale (VAS), registration 0 (=no pain)-100 (=worst pain), where In the minimal clinically significant change has been estimated as 11 points on a 100-point scale patients with rheumatoid arthritis, the minimal clinically significant change has been estimated as 1.1 points on an 11-point scale (or 11 points on a 100-point scale)
Change in Patient-reported pain | 12 months compared to baseline and 6 months
  Visual Analog Scale (VAS) registration 0 (=no pain)-100 (=worst pain), where In the minimal clinically significant change has been estimated as 11 points on a 100-point scale
Difference in T2 (transverse relaxation time) | 6 months compared to baseline
  MRI can characterize tissue by two different relaxation times, T1 and T2
Difference in T2 (transverse relaxation time) | 12 months compared to baseline and 6 months
  MRI can characterize tissue by two different relaxation times, T1 and T2

SECONDARY OUTCOMES:
Change in clinical outcomes (Standing inspection) | 6 months compared to baseline
  Normal spine curvature (yes/no)
Change in clinical outcomes (Standing side-to-side symmetry) | 6 months compared to baseline
  Standing side-to-side symmetry (yes/no)
Change in Clinical outcomes (Muscle hypotrophy) | 6 months compared to baseline
  Muscle hypotrophy (yes/no)
Change in Clinical outcomes (Walking on heels) | 6 months compared to baseline
  Ability to walk on heels (yes/no)
Change in Clinical outcomes (Walking on toes) | 6 months compared to baseline
  Ability to walk on toes (yes/no)
Change in Clinical outcomes (Standing inspection) | 12 months compared to baseline and 6 months
  Normal spine curvature (yes/no)
Change in Clinical outcomes (Standing side-to-side symmetry) | 12 months compared to baseline and 6 months
  Standing side-to-side symmetry (yes/no)
Change in Clinical outcomes (Muscle hypotrophy) | 12 months compared to baseline and 6 months
  Muscle hypotrophy (yes/no)
Change in Clinical outcomes (Walking on heels) | 12 months compared to baseline and 6 months
  Ability to walk on heels (yes/no)
Change in Clinical outcomes (Walking on toes) | 12 months compared to baseline and 6 months
  Ability to walk on toes (yes/no)
Change in Functional tests (Sit-to-stand test) | 6 months compared to baseline
  Sit-to-stand test (number of rises during 30 sec)
Change in Functional tests (Prone-bridge test) | 6 months compared to baseline
  Prone-bridge test (total sec)
Change in Functional tests (Åstrand ergometer test) | 6 months compared to baseline
  Åstrand ergometer test (estimated VO2-max, a measure of the maximum amount of oxygen your body can utilize during exercise)
Change in Functional tests (Sit-to-stand test) | 12 months compared to baseline and 6 months
  Sit-to-stand test (number of rises during 30 sec)
Change in Functional tests (Prone-bridge test) | 12 months compared to baseline and 6 months
  Prone-bridge test (total sec)
Change in Functional tests (Åstrand ergometer test) | 12 months compared to baseline and 6 months
  Åstrand ergometer test (estimated VO2-max)
Change in PROM (Standardized National standardized questions on physical activity) | 6 months compared to baseline
  Standardized National standardized questions on physical activity (grading activity in minutes/week).
Change in PROM (Oswestry Low Back Disability Index) | 6 months compared to baseline
  Oswestry Low Back Disability Index (0-4 No disability, 5-14 Mild disability, 15-24, Moderate disability, 25-34 Severe disability).
Change in PROM (Hospital Anxiety and Depression Scale (HAD)) | 6 months compared to baseline
  Hospital Anxiety and Depression Scale (HAD) 0-7 = Normal, 8-10 = Borderline abnormal, 11-21 = Abnormal).
Change in PROM (The 5-level EQ-5D version (EQ-5D-5L)) | 6 months compared to baseline
  The 5-level EQ-5D version (EQ-5D-5L) according to EuroQol Group The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in PROM (Tampa Scale of Kinesiophobia (TSK)) | 6 months compared to baseline
  Tampa Scale of Kinesiophobia (TSK) is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Change in PROM (Generalized Self-Efficacy Scale (GSES)) | 6 months compared to baseline
  Generalized Self-Efficacy Scale (GSES), a 10 item self-report measure of self-efficacy, with a higher score indicating more self-efficacy.
Change in PROM (Standardized National standardized questions on physical activity) | 12 months compared to baseline and 6 months
  Standardized National standardized questions on physical activity (grading activity in minutes/week).
Change in PROM (Oswestry Low Back Disability Index) | 12 months compared to baseline and 6 months
  Oswestry Low Back Disability Index (0-4 No disability, 5-14 Mild disability, 15-24, Moderate disability, 25-34 Severe disability).
Change in PROM (Hospital Anxiety and Depression Scale (HAD)) | 12 months compared to baseline and 6 months
  Hospital Anxiety and Depression Scale (HAD) 0-7 = Normal, 8-10 = Borderline abnormal, 11-21 = Abnormal).
Change in PROM (The 5-level EQ-5D version (EQ-5D-5L)) | 12 months compared to baseline and 6 months
  The 5-level EQ-5D version (EQ-5D-5L) according to EuroQol Group The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in PROM (Tampa Scale of Kinesiophobia (TSK)) | 12 months compared to baseline and 6 months
  Tampa Scale of Kinesiophobia (TSK) is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Change in PROM (Generalized Self-Efficacy Scale (GSES)) | 12 months compared to baseline and 6 months
  Generalized Self-Efficacy Scale (GSES), a 10 item self-report measure of self-efficacy, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ninni IE Sernert, PhD, Study Director — Göteborg University; Kerstin Lagerstrand, PhD, Study Chair — Göteborg University; Helena Brisby, PhD, Study Chair — Göteborg University; Hanna Hebelka Bolminger, PhD, Study Chair — Göteborg University
Locations (1):
- Ninni Sernert, Vänersborg, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT05679167/Prot_000.pdf